CLINICAL TRIAL: NCT06790576
Title: Optimizing Transcranial Magnetic Stimulation for Stimulant Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2024-32713
Record Dates: First submitted 2025-01-02; First posted 2025-01-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stimulant Use Disorder
Keywords: TMS; MRI

STUDY DESIGN:
Intervention Model Description: Three randomized groups for type of TMS stimulation (random, peak, and trough), triple-blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Participants assigned to closed-loop-peak
  Interventions: Other: closed-loop-peak
- Group 2 (Experimental): Participants assigned to open-loop
  Interventions: Other: Open-loop
- Group 3 (Experimental): Participants assigned to closed-loop-trough
  Interventions: Other: closed-loop-trough

INTERVENTIONS:
Other: closed-loop-peak — With single pulse TMS stimulation at F3 based on 10-20 EEG system, TMS evoked potentials (TEPs) will be collected under three TMS synchronization conditions: closed-loop-peak (each pulse synchronized to person's peak of theta waveform)
  Arms: Group 1
Other: Open-loop — With single pulse TMS stimulation at F3 based on 10-20 EEG system, TMS evoked potentials (TEPs) will be collected under three TMS synchronization conditions: open-loop (TMS pulse delivered without regard to EEG)
  Arms: Group 2
Other: closed-loop-trough — With single pulse TMS stimulation at F3 based on 10-20 EEG system, TMS evoked potentials (TEPs) will be collected under three TMS synchronization conditions: closed-loop-trough (each pulse synchronized to trough of theta waveform)
  Arms: Group 3

SUMMARY:
The study will recruit 50 adults with stimulant use disorder currently in treatment and abstinent for at least 2 weeks. The study will also recruit up to 10 healthy controls (adults without StUD) for initial study configuration. The study will consist of five steps that are expected to be completed over two lab visits.

Step 1: The 3T MRI scan will provide accurate prefrontal cortex anatomy for using neuronavigation for TMS. In addition, the study will use an analysis of resting fMRI connectivity to determine the location in the left DLPFC that has the maximum connectivity with the incentive-salience network.

Step 2: The study will use the data collected at the MRI to select the individual TMS location. EEG will be used to collect TEPs in response to single pulse TMS at the left DLPFC. Participants will then be randomized to one of three conditions: A) TMS unsynchronized with EEG, B) TMS synchronized with EEG theta frequency trough, and C) TMS synchronized with EEG theta frequency peak. The stimulation will be applied with an intensity of up to 120% of the resting motor threshold (which is a safe and common practice; Rossi et al., 2021). The intensity can be decreased for individual participants.

Step 3: Following randomization, the study will administer a pre-iTBS assessment.

Step 4: The study will compare brain and behavioral responses before and after the iTBS session with TMS and EEG synchronization as assigned by their randomized group.

Step 5: The study will administer a post-iTBS assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to provide consent and comply with all study procedures.
* Meets Diagnostic and Statistical Manual of Mental Disorders criteria for StUD (As assessed by MINI and self-report; Participants may have current comorbid drug use, but primary diagnosis must be StUD; does not apply to healthy control participants).
* At least 2 weeks of abstinence from substance use (other than caffeine or nicotine).
* Intention to remain in an addiction treatment program until intervention completion (does not apply to healthy control participants).
* Confident level of English language proficiency.

Exclusion Criteria:

* Any organic brain disorder (e.g. TBI, stroke).
* Head injury resulting in skull fracture or loss of consciousness exceeding 30 minutes.
* TMS contraindication (history of seizures, metallic cranial plates/screws or implanted device).
* MRI contraindications (unapproved metallic implants, pacemakers or any other implanted electrical device, shrapnel, metallic braces, non-removable body piercings, pregnancy, breathing or movement disorder, claustrophobia).
* Any psychotic disorder (Participants with other treated and stable psychiatric disorders will be included).
* Presence of a condition that would render study measures impossible to administer or interpret.
* Primary current substance use disorder diagnosis on a substance other than stimulants or cocaine, except for caffeine or nicotine.
* Greater than 9 months abstinence from substance use (does not apply to healthy control participants).
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
TEP individual response | 2 hours
  Use TMS-evoked potentials (TEPs) to assess individual response to three TMS-EEG synchronization methods: random, peak, and trough.
Cognitive response | Measured immediately after the iTBS
  Investigate the CSST task cognitive response to three TMS-EEG synchronization approaches during intermittent Theta Burst Stimulation (iTBS).

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States